CLINICAL TRIAL: NCT05407168
Title: Improving Decision-Making Encounters in Lung Cancer (I DECide) II: A Randomized Control Trial Of A Low-Literacy Conversation Tool
Brief Title: Improving Decision-Making Encounters in Lung Cancer Using a Low-Literacy Conversation Tool
Acronym: iDECIDE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other); American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Donald R Sullivan, MD, MA, MCR, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00023160; NCI-2021-09819 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00023160 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-10-05; First posted 2022-06-07 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Health Promotion; Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (decision aid) (Experimental): Patients review decision aid.
  Interventions: Other: Health Promotion and Education; Other: Questionnaire Administration
- Group II (standard of care) (Active Comparator): Patients receive standard of care.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Group II (standard of care)
Other: Health Promotion and Education — View decision aid
  Arms: Group I (decision aid)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the effectiveness of a conversation tool on patient-centered health and decision-making outcomes in patients with lung cancer making treatment decisions. This research is being conducted to help doctors understand the information patients need to participate in shared decision-making about their lung cancer treatment options. The focus of this research is to study how patients choose lung cancer treatment options and the information needed to make that choice, with a focus on patients with lower health literacy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Conduct a randomized, controlled trial evaluating the efficacy of a conversation tool on patient-centered health and decision-making outcomes among patients making lung cancer treatment decisions. A subset of participants from control and intervention groups will also have their clinic conversations with providers recorded II. Conduct in-depth, semi-structured qualitative audio or video recorded interviews among a subset of Aim 1 participants.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients review decision aid.

GROUP II: Patients receive standard of care.

After completion of study intervention, patients are followed up at 2 weeks, 3 months, and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* AIM 1: Suspected lung cancer
* AIM 1: English fluency
* AIM 1: > 6-month life expectancy
* AIM 1: Score of ≥ 3 on the cognitive impairment screener
* AIM 2 PARTICIPANTS: Participation in Aim 1
* AIM 2 CLINICIANS: Discussing lung cancer treatment decisions with Aim 1 participants

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Decision Conflict | Up to 6 months
  Will be assessed using the Decisional Conflict Scale, which contains 16 items. Higher scores indicate higher decisional conflict.
Efficacy of a conversation tool on patients' knowledge of lung cancer | Up 6 months
  Will be assessed using nine questions from previously validated measures.
Satisfaction with Communication/Confidence in Decision | Up to 6 months
  Will be assessed using the 20-item COMRADE scale. Higher scores indicate better outcomes.
Self-Efficacy | Up to 6 months
  Will be assessed using the Decision Self-Efficacy Scale which contains 11 items. Higher scores indicate higher self-efficacy.

SECONDARY OUTCOMES:
FACT-L | Up to 6 months.
  Quality of Life will be assessed by the Functional Assessment of Cancer Therapy -- Lung scale. This scale has 27 items. Higher scores indicate higher quality of life.
Depression/Anxiety | Up to 6 months
  Will be assessed using the 4 item Patient Health Questionnaire for Anxiety and Depression scale. Scores greater than or equal to 3 on the first two questions suggest anxiety, and scores greater than or equal to 3 on the last two questions suggest depression.
Participation in Decision-Making | Up to 6 months
  Will be assessed using the 2-item Control Preferences Scale. Answers of 1 or 2 on both items are categorized as "patient controlled", answers of 3 are categorized as "shared", and answers of 4 or 5 are categorized as "physician-controlled."
Decision Regret | Up to 6 months
  Will be assessed using the 5-item Decision Regret Scale. Higher scores indicate high regret.
Quality of Communication | Up to 6 months
  Will be assessed using the ~30 item Patient Assessment of cancer Communication Experiences scale. Higher scores indicate higher perceived quality of communication.
Number of Palliative Care Referrals | Up to 6 months
  Will be assessed by conducting chart review
Treatment Decision-Making Concordance | Up to 6 months
  Will be assessed by observing the treatment received and the treatment most aligned with responses to the conversation tool. If the treatment received is the same treatment the patient preferred according to the conversation tool, the treatment decision will be considered concordant.
Acceptability | Up to 6 months
  Will be assessed using the Ottawa Acceptability scale for patients in the intervention group only.

CONTACTS AND LOCATIONS:
Overall Officials: Donald R Sullivan, MD, MA, MCR, Principal Investigator — OHSU Knight Cancer Institute
Locations (4):
- United States (4):
  - Hillsboro Medical Center, Hillsboro, Oregon
  - Adventist Health Portland, Portland, Oregon
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon

REFERENCES:
- [Derived] Disher N, Dieckmann NF, Case JR, Rubim F, Eden KB, Golden SE, Matlock DD, Coleman C, Lyons KS, Saha S, Slatore CG, Vranas KC, Sullivan DR. Improving lung cancer decision-making using a conversation tool (iDECIDE): a stepped wedge pragmatic clinical trial. Future Oncol. 2025 Apr;21(9):1045-1056. doi: 10.1080/14796694.2025.2475733. Epub 2025 Mar 18. PMID 40098532